CLINICAL TRIAL: NCT02314338
Title: The Short Physical Performance Battery in COPD - Possible Impact of a Pulmonary Rehabilitation Program and Relationships to Other Physical Performance Measures, Symptoms, and Quality of Life.
Brief Title: The Short Physical Performance Battery in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REK2014/1499
Record Dates: First submitted 2014-11-27; First posted 2014-12-11 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary rehabilitation (Experimental): Multi-disciplinary pulmonary rehabilitation
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — In-patient pulmonary rehabilitation including individualized exercise prescription, group based exercise training, education, individual sessions with a multi professional health care team

SUMMARY:
Patients with COPD often have limitations to physical performance. There are several tests for evaluating physical performance, unfortunately many of them can be time consuming and require specialized equipment an substantial space. Short physical performance battery is a simple test that requires little resources and can be performed both at institutions and in the homes of patients. SPPB has high predictive abilities in identifying older adults at greater risk for mortality, nursing home admission, hospitalization, and incidence of disability. The investigators would like to evaluate possible changes in the SPPB score after a 4-week rehabilitation program. The investigators would also like to look at possible relationships between the SPPB and other physical performance measures, dyspnea, anxiety, depression, fatigue, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with all stages of COPD
* Decision making capacity to provide informed written consent
* Ability to understand and complete the questionnaires

Exclusion Criteria:

* Exacerbation within the last four weeks
* Co-morbidities that limits the patient's physical performance more than COPD
* Any patient whom is deemed unsafe to exercise
* Patients tested on treadmill protocol 4 (i.e. Glittre testing protocol)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Short physical performance battery (SPPB) | Pre and posttest with 4 weeks in between
  SPPB is comprised of 3 tasks: a hierarchial standing balance test (side by side, semi-tandem and tandem), 4-m habitual gait speed, and 5 sit to stand from a chair. Each task is scored (based on time) from 0-4 Points (p) and then summarized into a total score of 0-12 p, where 12 p represents the highest performance.

SECONDARY OUTCOMES:
Lung function | 4 weeks
  spirometry and/or whole body plethysmography
6-minute walk test (6MWT) | 4 weeks
  The 6 MWT is a timed walk test. Participants are asked to walk as far as possible, in 6 minutes. Borg CR-10 score and SpO2 will be measured before, during and/or after the 6 MWT.
Borg category ratio-10 scale (Borg CR-10 scale) | 4 weeks
  The Borg CR-10 scale is a rating scale for self-reported symptoms, in this case dyspnea. 0 represents no symptoms and 10 the worst previously experienced symptoms.
Peripheral oxygenation level | 4 weeks
  Peripheral oxygenation level (SpO2) will be measured indirectly by pulse oximetry during the 6 MWT.
Bilateral leg press 1 repetition Maximum (RM) | 4 weeks
  1 RM bilateral leg press will be administered, after a brief warm-up, as a measure of leg strength. Starting position: Legs shoulder width apart and knee at 90 degrees angle.
Modified Medical Research Council Dyspnea Scale (MMRC) | 4 weeks
  A score from 0-4 is used to classify the impact of dyspnea on physical function in patients with COPD. 0 represents a person who suffers from dyspnea only with strenuous exercise. 4 is a person who are to breathless to leave the house, or breathless when dressing/undressing.
COPD assessment test (CAT) | 4 weeks
  CAT is a disease-specific quality of life questionnaire. It has 8-items and a total range of 0-40, where 40 represents more severe impact of COPD on a patient's life.
Hospital anxiety and depression scale (HADS) | 4 weeks
  14-item questionnaire for screening for anxiety and depression. Each item is scored from 0-3 and each person can have a score between 0-21 for either anxiety or depression.
Fatigue severity scale (FSS) | 4 weeks
  9- item scale that measures the impact of fatigue on a person's activities and lifestyle. Range 9-63. Higher score- greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Edvardsen, PhD, Principal Investigator — LHL-klinikkene Glittre
Locations (1):
- LHL-klinikkene Glittre, Hakadal, Norway

REFERENCES:
- [Derived] Larsson P, Borge CR, Nygren-Bonnier M, Lerdal A, Edvardsen A. An evaluation of the short physical performance battery following pulmonary rehabilitation in patients with chronic obstructive pulmonary disease. BMC Res Notes. 2018 Jun 4;11(1):348. doi: 10.1186/s13104-018-3458-7. PMID 29866200